CLINICAL TRIAL: NCT03917173
Title: Prophylactic Surgery Plus Hyperthermic Intraperitoneal Chemotherapy (HIPEC CO2) Versus Standard Surgery in Gastric Carcinoma at High Risk of Developing Peritoneal Carcinomatosis. Short and Long-term Outcomes Evaluation.A Collaborative Randomized Controlled Trial of: ACOI, FONDAZIONE AIOM, SIC, SICE, SICO. GOETH STUDY
Brief Title: Prophylactic Surgery Plus HIPEC With CO2 in Patients Affected by Gastric Carcinoma.GOETH Study
Acronym: GOETH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-GCC-7813; 2019-001478-27 (EudraCT Number)
Record Dates: First submitted 2019-04-02; First posted 2019-04-16 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Stomach Neoplasms
Keywords: gastric cancer; HIPEC CO2; Prophylactic surgery; hyperthermic intraperitoneal chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: This is a phase III randomized, multicenter study with two different arm:
  * experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin and cisplatin
  * comparator: standard surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Prophylactic surgery plus HIPEC CO2 performed with mitomycin and cisplatin
  Interventions: Procedure: Surgery plus HIPEC CO2
- Comparator (Active Comparator): Standard surgery
  Interventions: Procedure: Standard surgery

INTERVENTIONS:
Procedure: Surgery plus HIPEC CO2 — Prophylactic surgery plus HIPEC CO2 performed with mitomycin and cisplatin v
  Arms: Experimental
Procedure: Standard surgery — Standard surgery without HIPEC CO2
  Arms: Comparator

SUMMARY:
This is a phase III randomized, multicenter study with two different arm:

* experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin and cisplatin
* comparator: standard surgery

Adjuvant treatment after surgery is mandatory except for documented cases of non-eligibility in both arms.

Patient will be randomized in a 1:1 ratio. Randomization will be performed during surgery if the total resection of tumor will be reached according to center and neoadjuvant chemotherapy as stratification variables.

DETAILED DESCRIPTION:
This is a phase III randomized, multicenter study with two different arm:

* experimental: prophylactic surgery plus HIPEC CO2 performed with mitomycin and cisplatin
* comparator: standard surgery Adjuvant treatment after surgery is mandatory except for documented cases of non-eligibility.

Patient will be randomized in a 1:1 ratio. Randomization will be performed during surgery if the total resection of tumor will be reached according to center and neoadjuvant chemotherapy as stratification variables.

The primary objective of the study is to compare the efficacy of prophylactic surgery (radical gastric resection, appendectomy, round ligament of the liver resection and bilateral adnexectomy) plus HIPEC CO2 versus standard surgery in terms of disease free survival (DFS).

Patients affected by gastric carcinoma at high risk of developing peritoneal carcinomatosis will be randomized in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically documented gastric carcinoma (diffuse/intestinal histotype) eligibile for R0.

   1. Presurgical or intraoperative stage T3-T4 N0-N+ primary tumour (TNM 8 th).
   2. Urgent presentation: perforation without purulent generalized peritonitis
   3. Positive cytology of peritoneal fluid (if previously obtained)
2. Age ≥ 18 years and ≤75 years.
3. Written informed consent.

Exclusion Criteria:

1. Gastroesophageal Junction (GEJ) cancer
2. Distant metastatic disease (even if limited and completely resected)
3. Peritoneal carcinomatosis
4. History of tumor diagnosed in the 3 years before entering the study, except for topical and healed pathologies that do not need further treatment (e.g. non-melanoma skin carcinomas, superficial bladder carcinomas or in situ carcinoma of the breast or cervix).
5. Psychological, family or social conditions which may negatively affect the treatment and follow-up protocol.
6. Poor general conditions (ECOG > 2).
7. Impaired cardiac function (history of congestive heart failure or FE <40%). Clinically significant cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrolment), unstable angina, congestive heart failure (New York Heart Association Classification Class > II) or serious uncontrolled cardiac Arrhythmia requiring medication
8. Impaired renal function (creatinine> 1.5 upper limit of normal or creatinine clearance <60 mL / min).
9. Impaired hepatic function (AST, ALT >2.5 upper limit of normal, bilirubin > 1.5 upper limit of normal).
10. Impaired hematopoietic function (leucocytes <4000 / mm3, neutrophils <1500 / mm 3, platelets <100000 / mm3).
11. Impaired pulmonary function (presence of COPD or other pulmonary restrictive conditions with FEV1 <50% or DLCO <40% of normal age value).
12. History or presence of other disease, metabolic dysfunction, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of HIPEC or chemotherapy or patient at high risk from treatment complications.
13. Pregnancy.
14. Krukenberg tumor
15. Refusal to join the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  The primary efficacy endpoint is DFS defined as the time from randomization to the date of first local relapse or distant relapse or peritoneal carcinomatosis or death for any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival | This outcome measure will be assessed approximately 3 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Overall Survival (OS) defined as the time from randomization to the death for any cause
Local recurrence free survival | This outcome measure will be assessed approximately 3 years after the last patient enrolled, at the same time points of the Primary Endpoint
  Local recurrence free survival (LRFS) defined as the time from randomization defined as the time from randomization to the date of first local relapse, peritoneal carcinomatosis or death for any cause, whichever comes first.
morbidity evaluated during and after surgery | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  morbidity evaluated during and after surgery graded according to the NCI-CTAE version 4.03 for AE related to chemotherapy and according to Clavien Dindo for surgery complications
post-surgery complication | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  number of post-surgery complication
duration of surgery | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  timing of surgery
length of hospitalization | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  duration of hospitalization
mortality at 30 and 90 days from surgery | This outcome measure will be assessed at 30 and 90 days from surgery
  mortality at 30 and 90 days from surgery
patients performing the adjuvant chemotherapy. | This outcome measure will be assessed approximately 3 years after the last patient enrolled
  number of patients performing the adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Di Giorgio, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (12):
- Italy (12):
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - AO Santa Croce e Carle, Cuneo
  - ULLS1 1 Dolomiti - Ospedale di Feltre, Feltre
  - Policlinico di Milano, Milan
  - A.O.R.N. A.Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Ospedale Evangelico Betania, Napoli
  - Azienda Ospedaliera S. Camillo Forlanini, Roma
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs Universita' Cattolica Del Sacro Cuore, Roma
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Giorgio A, Gerardi C, Abatini C, Melotti G, Bonavina L, Torri V, Santullo F, Garattini S, De Luca M, Rulli E, Rulli E, Pacelli F; GOETH Investigators. Prophylactic surgery plus hyperthermic intraperitoneal chemotherapy (HIPEC CO2) versus standard surgery for gastric carcinoma at high risk of peritoneal carcinomatosis: short and long-term outcomes (GOETH STUDY)-a collaborative randomized controlled trial by ACOI, FONDAZIONE AIOM, SIC, SICE, and SICO. Trials. 2022 Dec 1;23(1):969. doi: 10.1186/s13063-022-06880-y. PMID 36457115